CLINICAL TRIAL: NCT05902715
Title: The Socket Shield Technique: Stability of the Buccal Peri-implant Bone After Partial Root Removal - a Prospective Cohort Study of 20 Patients, With 18 Months Follow-up
Brief Title: The Socket Shield Technique, a Prospective Cohort Study of 20 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Ana CASTRO SARDA, Clinical professor, head of periodontology department, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S59423
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2023-06

CONDITIONS: Peri-implant Health
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- oral implant placement with socket shield technique (Experimental): cohort of 20 patients in need of tooth replacement with oral implant
  Interventions: Device: oral implant placement with socket shield technique

INTERVENTIONS:
Device: oral implant placement with socket shield technique — tooth is split in socket shield configuration, implant is immediately placed

SUMMARY:
23 implants with socket shield were followed for 18 months. buccal bone thickness and survival rates registered.

DETAILED DESCRIPTION:
Aims: This study aims to collect data on implant survival, bone volume maintenance, and complications associated with the socket shield technique.

Materials & methods: The study involved the placement of 23 implants using the socket shield technique in 20 patients. AstraTech EV implants were used, and no bone substitutes or connective tissue grafts were applied. Patients were monitored for 18 months, recording implant survival, volumetric bone analysis on CBCT scans, interproximal bone levels, bone sounding, pink esthetic scores, and complications. Prosthetic procedures were also described, including temporary and final restorations.

ELIGIBILITY:
Inclusion Criteria:

* • Hopeless teeth suitable for immediate implant placement

  * Only single-rooted teeth in the maxilla
  * Intact buccal and palatal bone plate
  * Intact buccal root portion
  * Any periodontal phenotype (thin, thick)

Exclusion Criteria:

* • Horizontal root fracture below bone level

  * Smoking
  * Systemic pathology influencing bone healing
  * Active periodontal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
buccal bone thickness | 18 months
  thickness as measured on cbct scan

SECONDARY OUTCOMES:
Cumulative survival rate | 18 months
  implant survival

CONTACTS AND LOCATIONS:
Overall Officials: Rutger Dhondt, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No